CLINICAL TRIAL: NCT00163358
Title: Efficacy of Ciclesonide and of a Fixed Combination With Fluticasone Propionate and Salmeterol Versus Placebo on Long-term Asthma Control
Brief Title: Efficacy of Ciclesonide vs Fixed Combination of Fluticasone Propionate/Salmeterol vs Placebo in Patients With Mild Persistent Asthma (12 to 75 y) (BY9010/M1-132)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-132
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Fluticasone propionate; Salmeterol
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the study is to compare the efficacy of ciclesonide versus fixed combination of fluticasone propionate/salmeterol versus placebo, on long-term asthma control in patients with mild persistent asthma. The study duration consists of a baseline period (2 weeks) and a treatment period (12 months). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Clinical diagnosis of mild persistent asthma
* Pre-treatment with SABAs only
* FEV1 ≥80% predicted
* Good health with the exception of asthma

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* COPD (chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in pulmonary function
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception
* Current smokers ≥10 pack-years and ex-smokers with ≥10 pack-years

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 630
Dates: Start 2003-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
time until the first severe asthma exacerbation occurs
number of poorly controlled asthma days.

SECONDARY OUTCOMES:
percentage of days with asthma control
percentage of days with asthma symptoms
percentage of nocturnal awakenings due to asthma
asthma symptom score
number of inhalations of rescue medication
proportion of patients with severe asthma exacerbations
differences in morning PEF from diary
differences in FEV1 and FVC from spirometry
blood eosinophils
AQLQ(S)
health economic data
vital signs
laboratory work-up
adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (97):
- Australia (16):
  - Altana Pharma/Nycomed, Adelaide South Australia
  - Altana Pharma/Nycomed, Auchenflower
  - Altana Pharma/Nycomed, Bracken Ridge
  - Altana Pharma/Nycomed, Burwood
  - Altana Pharma/Nycomed, Camperdown
  - Altana Pharma/Nycomed, Carina Heights
  - Altana Pharma/Nycomed, Clayton
  - Altana Pharma/Nycomed, Concord
  - Altana Pharma/Nycomed, Geelong
  - Altana Pharma/Nycomed, Inala
  - Altana Pharma/Nycomed, Kippa-Ring
  - Altana Pharma/Nycomed, Nedlands
  - Altana Pharma/Nycomed, Rosebud
  - Altana Pharma/Nycomed, South Brisbane
  - Altana Pharma/Nycomed, Toorak Gardens
  - Altana Pharma/Nycomed, Wayville
- Canada (24):
  - Altana Pharma/Nycomed, Beaconsfield, QC
  - Altana Pharma/Nycomed, Coquitlam
  - Altana Pharma/Nycomed, Coquitlam, BC
  - Altana Pharma/Nycomed, Corner Brook
  - Altana Pharma/Nycomed, Cowansville
  - Altana Pharma/Nycomed, Kingston, Ontario
  - Altana Pharma/Nycomed, Langley BC
  - Altana Pharma/Nycomed, Laval
  - Altana Pharma/Nycomed, Les Saules, QC
  - Altana Pharma/Nycomed, Longueuil, PQ
  - Altana Pharma/Nycomed, Montreal
  - Altana Pharma/Nycomed, Montreal, PQ
  - Altana Pharma/Nycomed, North Bay
  - Altana Pharma/Nycomed, North York
  - Altana Pharma/Nycomed, Ottawa
  - Altana Pharma/Nycomed, Penticton, BC
  - Altana Pharma/Nycomed, Québec
  - Altana Pharma/Nycomed, Saint John
  - Altana Pharma/Nycomed, Sainte-Foy, Quebec
  - Altana Pharma/Nycomed, Saskatoon, SK
  - Altana Pharma/Nycomed, St. John's
  - Altana Pharma/Nycomed, Ste-Foy PQ
  - Altana Pharma/Nycomed, Toronto
  - Altana Pharma/Nycomed, Toronto on
- Czechia (17):
  - Altana Pharma/Nycomed, Beroun
  - Altana Pharma/Nycomed, Cvikov
  - Altana Pharma/Nycomed, Česká Lípa
  - Altana Pharma/Nycomed, Havlickuv
  - Altana Pharma/Nycomed, Jihlava
  - Altana Pharma/Nycomed, Jindřichův Hradec
  - Altana Pharma/Nycomed, Karlovy Vary
  - Altana Pharma/Nycomed, Kladno
  - Altana Pharma/Nycomed, Kutná Hora
  - Altana Pharma/Nycomed, Ostrava-Marián.Hory
  - Altana Pharma/Nycomed, Prague
  - Altana Pharma/Nycomed, Pribram VI
  - Altana Pharma/Nycomed, Príbram VIII
  - Altana Pharma/Nycomed, Rokycany
  - Altana Pharma/Nycomed, Strakonice
  - Altana Pharma/Nycomed, Trutnov
  - Altana Pharma/Nycomed, Ústí nad Labem
- Hungary (7):
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Budapest XI
  - Altana Pharma/Nycomed, Budapet
  - Altana Pharma/Nycomed, Kecskemét
  - Altana Pharma/Nycomed, Nyíregyháza
  - Altana Pharma/Nycomed, Szarvas
  - Altana Pharma/Nycomed, Tatabánya
- Poland (6):
  - Altana Pharma/Nycomed, Bydgoszcz
  - Altana Pharma/Nycomed, Lodz
  - Altana Pharma/Nycomed, Lódz'
  - Altana Pharma/Nycomed, Rzeszów
  - Altana Pharma/Nycomed, Warsaw
  - Altana Pharma/Nycomed, Wroclaw
- South Africa (14):
  - Altana Pharma/Nycomed, Arcadia, Pretoria
  - Altana Pharma/Nycomed, Bellville, Cape Town
  - Altana Pharma/Nycomed, Berea, Durban
  - Altana Pharma/Nycomed, Bloemfontein
  - Altana Pharma/Nycomed, Cape Town
  - Altana Pharma/Nycomed, Centurion, Pretoria
  - Altana Pharma/Nycomed, Daveyton
  - Altana Pharma/Nycomed, Durban, Amanzimtoti
  - Altana Pharma/Nycomed, George
  - Altana Pharma/Nycomed, Midrand
  - Altana Pharma/Nycomed, Mowbray, Cape Town
  - Altana Pharma/Nycomed, Paarl
  - Altana Pharma/Nycomed, Panorama / RSA-Cape Town
  - Altana Pharma/Nycomed, Pretoria
- Spain (13):
  - Altana Pharma/Nycomed, Alcorcón (Madrid)
  - Altana Pharma/Nycomed, Alicante
  - Altana Pharma/Nycomed, Barcelona
  - Altana Pharma/Nycomed, Campdevanol (Girona)
  - Altana Pharma/Nycomed, Elda (Alicante)
  - Altana Pharma/Nycomed, Guadalajara
  - Altana Pharma/Nycomed, Leganes (Madrid)
  - Altana Pharma/Nycomed, Palma de Mallorca
  - Altana Pharma/Nycomed, Peralada (Girona)
  - Altana Pharma/Nycomed, Petrer (Alicante)
  - Altana Pharma/Nycomed, San Vicente Del Raspeig (Alicante)
  - Altana Pharma/Nycomed, Santiago de Compostela
  - Altana Pharma/Nycomed, Valencia

REFERENCES:
- [Derived] Postma DS, O'Byrne PM, Pedersen S. Comparison of the effect of low-dose ciclesonide and fixed-dose fluticasone propionate and salmeterol combination on long-term asthma control. Chest. 2011 Feb;139(2):311-318. doi: 10.1378/chest.09-1735. Epub 2010 Nov 18. PMID 21088114
- See also: BY9010-MI-132-RDS-2007-02-12.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4520&filename=BY9010-MI-132-RDS-2007-02-12.pdf